CLINICAL TRIAL: NCT05639894
Title: A Phase I/IIa, Randomized, Placebo-controlled Multi-arm Dose-finding Study to Evaluate the Safety and Immunogenicity of a RSV Vaccine Candidate in Adult Participants 18 to 50 Years of Age in Phase I, and 60 Years and Older in Phase IIa
Brief Title: Study of a Respiratory Syncytial Virus Candidate Encapsulated in a Lipid Nanoparticle Based Formulation in Adults Aged 18 to 50 Years and 60 Years and Older
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VAE00010; U1111-1271-1514 (Registry Identifier: ICTRP); 2023-505343-40 (Registry Identifier: CTIS)
Record Dates: First submitted 2022-11-17; First posted 2022-12-07 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Respiratory Syncytial Virus Immunization

STUDY DESIGN:
Intervention Model Description: Sequential (Phase I)/ parallel (Phase IIa)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sentinel Cohort: single-blind
  * Investigators, study staff who conduct the safety assessment, and the participant will not know which study intervention is administered
  * Sponsor study staff and study staff preparing/administering the study interventions and not involved with the safety evaluation will know which study intervention is administered Main and Booster Cohorts in Stage 1 and Stage 2: Modified double-blind
  * Investigators, study staff who conduct the safety assessment, and the participant will not know which study intervention is administered
  * Only the study staff who prepare and administer the study intervention and are not involved with the safety evaluation will know which study intervention is administered
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (10):
- Group 1: Sentinel and Main Cohorts (Stage 1) (Experimental): 1 injection of RSV vaccine candidate (Dose A) via intramuscular injection
  Interventions: Biological: RSV vaccine candiate formulation 1
- Group 2: Sentinel and Main Cohorts (Stage 1) (Experimental): 1 injection of RSV vaccine candidate (Dose A) via intramuscular injection
  Interventions: Biological: RSV vaccine candidate formulation 2
- Group 3: Sentinel and Main Cohorts (Stage 1) (Experimental): 1 injection of RSV vaccine candidate (Dose B) via intramuscular injection
  Interventions: Biological: RSV vaccine candiate formulation 1
- Group 4: Sentinel and Main Cohorts (Stage 1) (Experimental): 1 injection of RSV vaccine candidate (Dose B) via intramuscular injection
  Interventions: Biological: RSV vaccine candidate formulation 2
- Group 5: Sentinel and Main Cohorts (Stage 1) (Experimental): 1 injection of RSV vaccine candidate (Dose C) via intramuscular injection
  Interventions: Biological: RSV vaccine candiate formulation 1
- Group 6: Sentinel and Main Cohorts (Stage 1) (Experimental): 1 injection of RSV vaccine candidate (Dose C) via intramuscular injection
  Interventions: Biological: RSV vaccine candidate formulation 2
- Group 7: Main, Sentinel and Booster Cohorts (Stage 1) (Placebo Comparator): 1 injection of placebo via intramuscular injection
  Interventions: Other: Placebo
- Group 0: Phase IIa/Dose-ranging (Stage 2) (Experimental): 1 injection of RSV vaccine candidate (Dose A) via intramuscular injection
  Interventions: Biological: RSV vaccine candiate formulation 1
- Group 1: Phase IIa/Dose-ranging (Stage 2) (Experimental): 1 injection of RSV vaccine candidate (Dose B) via intramuscular injection
  Interventions: Biological: RSV vaccine candidate formulation 2
- Group 2: Phase 11a/Dose-ranging (Stage 2) (Placebo Comparator): 1 injection of placebo via intramuscular injection
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: RSV vaccine candiate formulation 1 — Pharmaceutical Form: Liquid frozen solution in a vial Route of Administration: Intramuscular injection
  Arms: Group 0: Phase IIa/Dose-ranging (Stage 2); Group 1: Sentinel and Main Cohorts (Stage 1); Group 3: Sentinel and Main Cohorts (Stage 1); Group 5: Sentinel and Main Cohorts (Stage 1)
Biological: RSV vaccine candidate formulation 2 — Pharmaceutical Form: Liquid frozen solution in a vial Route of Administration: Intramuscular injection
  Arms: Group 1: Phase IIa/Dose-ranging (Stage 2); Group 2: Sentinel and Main Cohorts (Stage 1); Group 4: Sentinel and Main Cohorts (Stage 1); Group 6: Sentinel and Main Cohorts (Stage 1)
Other: Placebo — Pharmaceutical Form: Liquid Route of Administration: Intramuscular injection
  Arms: Group 2: Phase 11a/Dose-ranging (Stage 2); Group 7: Main, Sentinel and Booster Cohorts (Stage 1)

SUMMARY:
Brief Summary of Stage 1:

The purpose Stage 1 (Phase I/IIa) is to assess the safety and immunogenicity of a single intramuscular (IM) injection of 3 dose-levels of an Respiratory Syncytial Virus (RSV) vaccine candidate formulated with 2 different lipid nanoparticles (LNPs) in healthy adult participants aged between 18 to 50 years, and 60 years and older. The primary objectives of this stage are to assess the safety and immunogenicity profiles across the dose-level groups (low, medium, and high doses) with 2 LNPs. This stage will evaluate the safety and immunogenicity of a booster vaccination administered 12 months after the primary vaccination in a subset of the study population.

Brief Summary of Stage 2:

The study also also incorporates a Stage 2 (Phase IIa, dose-ranging design) that includes adults aged 60 years and older to assess the safety and immunogenicity of different doses of RSV vaccine encapsulated in one of the LNPs. In the Phase IIa dose-ranging stage, eligible participants will be randomly assigned in a 1:1:1 ratio to receive a single IM administration of RSV vaccine candidate doses, or placebo. Multiple safety analyses will be performed, minimally at D07 and D28. Additional analyses may be performed as data are available.

DETAILED DESCRIPTION:
Stage 1:

The duration of each participant's participation is 12 months for the Sentinel and Main Cohorts, 24 months overall for the subset of participants enrolled in the Booster Cohort.

Treatment Duration:

* Sentinel Cohort: 1 intra-muscular (IM) injection. Participants will be followed for 12 months post-vaccination.
* Main Cohort: 1 IM injection. Participants will be followed for 12 months post-vaccination.
* Booster Cohort: 1 IM injection 12 months after the primary vaccination. Participants will be followed for 12 months after administration of the booster dose.

Stage 2:

The duration of each participant's participation is approximately 6 months.

Treatment Duration:

1 IM injection. Participants will be followed for approximately 6 months post vaccination

ELIGIBILITY:
Inclusion Criteria:

* Sentinel Cohort Stage 1: Aged 18 to 50 years on the day of inclusion
* Main Cohort Stage 1 and Stage 2: Aged 60 years or older on the day of inclusion

Stage 1 and Stage 2:

* Sentinel Cohort: A female participant is eligible to participate if she is not pregnant or breastfeeding and:

  * Is of non-childbearing potential. To be considered of non-childbearing potential, a female must be postmenopausal for at least 1 year or surgically sterile OR
  * Is of childbearing potential and agrees to use an effective contraceptive method or abstinence from at least 4 weeks prior to study intervention administration until at least 12 weeks after study intervention administration.
* Main and Booster Cohorts: A female participant is eligible to participate if she is not pregnant or breastfeeding and:

  * Is of non-childbearing potential. To be considered of non-childbearing potential, a female must be postmenopausal for at least 1 year or surgically sterile.
* Able to attend all scheduled visits and to comply with all study procedures
* Informed consent form has been signed and dated

Exclusion Criteria:

* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Known systemic hypersensitivity to any of the study intervention components (eg, polyethylene glycol, polysorbate); history of a life-threatening reaction to the study interventions used in the study or to a product containing any of the same substances; any allergic reaction (eg, anaphylaxis) after administration of mRNA COVID-19 vaccine
* History of RSV-associated illness, diagnosed clinically, serologically, or microbiologically in the last 12 months
* Previous history of myocarditis, pericarditis, and/or myopericarditis
* Thrombocytopenia or bleeding disorder, contraindicating IM injection based on investigator's judgment
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating intramuscular injection
* Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with study conduct or completion
* Alcohol, prescription drug, or substance abuse that, in the opinion of the investigator, might interfere with the study conduct or completion
* Receipt of any vaccine other than mRNA vaccine in the 4 weeks preceding any study intervention administration or planned receipt of any vaccine other than mRNA vaccine in the 4 weeks following any study intervention administration
* Receipt of any mRNA vaccine in the 60 days preceding any study intervention administration or planned receipt of any mRNA vaccine in the 60 days following any study intervention administration
* Previous vaccination against RSV with an investigational vaccine
* Receipt of immune globulins, blood, or blood-derived products in the past 3 months
* Receipt of oral or injectable antibiotic therapy within 72 hours prior to the first blood draw
* Participation at the time of study enrollment (or in the 4 weeks preceding the first study intervention administration) or planned participation during the present study period in another clinical study investigating a vaccine, drug, medical device, or medical procedure
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily
* Self-reported or documented human immunodeficiency virus (HIV) detected by any FDA-approved/validated test, hepatitis B virus surface antigen (HBsAg), hepatits B core antibodies (HBcAb), or hepatitis C virus antibodies (HCV Abs), or positive SARS-CoV-2 RT-PCR or antigen test
* Identified as an investigator or employee of the investigator or study center with direct involvement in the proposed study, or identified as an immediate family member (ie, parent, spouse, natural or adopted child) of the investigator or employee with direct involvement in the proposed study

The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 865 (Actual)
Dates: Start 2022-11-17 (Actual); Primary Completion 2025-05-02 (Actual); Study Completion 2025-05-02 (Actual)

PRIMARY OUTCOMES:
Presence of unsolicited systemic adverse events (AEs) | Within 30 minutes after vaccination
  Number of participants experienciing unsolicited systemic adverse events
Presence of solicited injection site or systemic reactions | Within 7 days after vaccination
  Number of participants reporting:
  * injection site reactions: pain, erythema and swelling
  * systemic reactions: fever, headache, malaise, myalgia, arthralgia and chills
Presence of unsolicited AEs | Within 28 days after vaccination
  Number of participants experiencing unsolicited AEs
Presence of medically attended adverse events (MAAEs) | Within 28 days after vaccination
  Number of participants experiencing MAAEs
Presence of serious adverse events (SAEs) | Month 12
  Number of participants experiencing SAEs
Presence of adverse events of special interest (AESIs) | Month 12
  Number of participants experiencing AESIs
Presence of out-of-range biological test results | Within 7 days after vaccination
  Number of participants with biological safety assessment values out of normal range (as per the laboratory performing the test)
Geometric Mean Titers (GMTs) of neutralizing antibody (nAb) titers pre-vaccination at Day 1 | Day 1
  Nab titers pre-vaccination
Geometric Mean Titers (GMTs) of neutralizing antibody (nAb) titers post-primary vaccination at Day 29 | Day 29
  Nab titers post-vaccination

SECONDARY OUTCOMES:
Presence of immediate unsolicited systemic AEs (Stage 1) | Within 30 minutes after vaccination
  Number of participants experiencing immediate unsolicitied systemic AEs
Presence of solicited injection site or systemic reactions post-booster vaccination (Stage 1) | Within 7 days after vaccination
  Number of participants reporting:
  * injection site reactions: pain, erythema and swelling
  * systemic reactions: fever, headache, malaise, myalgia, arthralgia and chills
Presence of unsolicited AEs post-booster vaccination (Stage 1) | Within 28 days after vaccination
  Number of participants experiencing unsolicited AEs
Presence of MAAEs (Stage 1) | Within 28 days after vaccination
  Number of participants experiencing MAAEs
Presence of serious adverse events (SAEs) post-booster vaccination (Stage 1) | Throughout the booster study, approximately 12 months
  Number of participants experiencing SAEs
Presence of adverse events of special interest post-booster vaccination (Stage 1) | Throughout the booster study, approximately 12 months
  Number of participants experiencing AESIs
Presence of out-of-range biological test results post-booster vaccination (Stage 1) | Within 7 days after vaccination
  Number of participants with biological safety assessment values out of normal range (as per the laboratory performing the test)
RSV-A serum nAb titers at pre-vaccination (D01) and 28 days post- primary vaccination (D29) (Stage 1) | Day 1, Day 29, Month 3, Month 6 and Month 12
  RSV-A serum nAb titers at pre-vaccination (D01), 28 days (D29), and 3, 6, and 12 months post-primary vaccination
GMTs of serum anti-F immunoglobulin G (IgG) antibody (Ab) titers post-primary vaccination (Stage 1) | Day 1, Day 29, Month 3, Month 6 and Month 12
  Serum anti-F IgG Ab titers at pre-vaccination (D01), 28 days (D29), and 3, 6, and 12 months post-primary vaccination
GMTs of RSV-A serum nAb post-booster vaccination (Stage 1) | Day 1, Day 29, Month 3, Month 6 and Month 12 post-booster
  RSV-A serum nAb titers at pre-booster vaccination, 28 days, and 3, 6, and 12 months post-booster vaccination
GMTs of serum anti-F IgG Ab titers post-booster vaccination (Stage 1) | Day 1, Day 29, Month 3, Month 6 and Month 12 post-booster
  Serum anti-F IgG Ab titers at pre-booster vaccination, 28 days, and 3, 6, and 12 months post- booster vaccination
GMTs of serum anti-F IgG Ab titers pre-vaccination (Stage 2) | Day 1
  Nab titers pre-primary vaccination
GMTs of serum anti-F IgG Ab titers post-vaccination (Stage 2) | Day 29
  Nab titers post-vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (33):
- United States (25):
  - Optimal Research Alabama Site Number : 8400032, Huntsville, Alabama
  - Aventiv Research Mesa Site Number : 8400020, Mesa, Arizona
  - CVS Health - Peoria Site Number : 8400042, Peoria, Arizona
  - CVS Health - Phoenix Site Number : 8400041, Phoenix, Arizona
  - Velocity Clinical Research - San Diego - ERN - PPDS Site Number : 8400010, La Mesa, California
  - Peninsula Research Associates Site Number : 8400013, Rolling Hills Estates, California
  - CVS Health - Thousand Oaks Site Number : 8400043, Thousand Oaks, California
  - Cenexel Research Centers of America Site Number : 8400024, Hollywood, Florida
  - Suncoast Research Associates, LLC Site Number : 8400003, Miami, Florida
  - Centricity Research - Georgia Site Number : 8400009, Rincon, Georgia
  - AES Peoria Site Number : 8400030, Peoria, Illinois
  - DM Clinical Research - Chicago Site Number : 8400027, River Forest, Illinois
  - Be Well Clinical Studies Site Number : 8400036, Lincoln, Nebraska
  - Velocity Clinical Research Site Number : 8400019, Cincinnati, Ohio
  - Velocity Clinical Research Site Number : 8400017, Cleveland, Ohio
  - Aventiv Research Columbus Site Number : 8400007, Columbus, Ohio
  - Lynn Institute of Norman Site Number : 8400023, Norman, Oklahoma
  - Velocity Clinical Research, Medford Site Number : 8400014, Medford, Oregon
  - Velocity Clinical Research - Providence Site Number : 8400006, East Greenwich, Rhode Island
  - Coastal Carolina Research Center Site Number : 8400015, North Charleston, South Carolina
  - DM Clinical Research - CyFair Site Number : 8400025, Houston, Texas
  - Be Well Clinical Studies -Round Rock Site Number : 8400038, Round Rock, Texas
  - IMA Clinical Research-San Antonio Site Number : 8400039, San Antonio, Texas
  - Martin Diagnostic Clinic Site Number : 8400026, Tomball, Texas
  - Velocity Clinical Research Site Number : 8400018, West Jordan, Utah
- Australia (3):
  - Investigational Site Number : 0360003, Botany, New South Wales
  - Investigational Site Number : 0360002, Camberwell, Victoria
  - Investigational Site Number : 0360001, Southport
- Puerto Rico (5):
  - Investigational Site Number : 6300004, Carolina
  - Investigational Site Number : 6300003, Guayama
  - Investigational Site Number : 6300005, Guaynabo
  - Investigational Site Number : 6300001, San Juan
  - Investigational Site Number : 6300002, San Juan

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org